CLINICAL TRIAL: NCT01256931
Title: Antibody Levels Against 2009 Influenza A H1N1 One Year After Vaccination With Pandemrix and 2010 Fluarix Booster in Organ Transplant Recipients.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Associate Professor Vanda Friman, Sahlgrenska University Hospital
Other Study IDs: MMV-305
Record Dates: First submitted 2010-12-07; First posted 2010-12-09 (Estimated); Last update posted 2010-12-09 (Estimated); Status verified 2010-12

CONDITIONS: Organ Transplantation
Keywords: 2009 H1N1 influenza vaccine, organ transplant patients,; booster with Fluarix

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- organ transplant patients
- healthy controls

SUMMARY:
Organ transplant patients who participated in a retrospective study and received 2009 Pandemrix vaccine during autumn 2009 are included in this study.

The main aim is to determine the H1N1 antibody levels one year after Pandemrix in comparison to healthy controls. The secondary aim is to examine the booster effect of 2010 Fluarix in patients and controls.Side effects to Fluarix vaccine are registered.

DETAILED DESCRIPTION:
Organ transplant patients and staff members of the Transplant Institute who were vaccinated 2009 and received 2 doses of 2009 H1N1 influenza vaccine (Pandemrix) will be asked to participate in the study.

Serum samples will be collected approximately one year after completed vaccination with Pandemrix and analysed for haemagglutination -inhibiting antibodies against H1N1.The frequency of individuals with remaining protective titers will be examined.

The same individuals will be vaccinated with Fluarix containing antigen from Influenza A California/7/2009(H1N1, A/Perth/16/2009 (H3N2) and B/Brisbane/60/2008. The booster effect will be measured one month later.

ELIGIBILITY:
Inclusion Criteria Cohort number 1: Organ transplant patients who were vaccinated with Pandemrix 2009 and written informed consent received

Cohort number 2: Staff members who were vaccinated with Pandemrix 2009 and written informed consent received

Exclusion Criteria:

Patients or controls who are allergic to formaldehyde, gentamycin sulphate or natrium deoxycholate or have other contraindications against to Fluarix vaccination.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Transplant patients at the out-patient clinical ward and staff members of the Transplant Institute, Sahlgrenska University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2010-12

PRIMARY OUTCOMES:
Frequency of individuals with remaining protective antibody titers against influenza H1N1 2009 one year after Pandemrix vaccination in organ transplant patients and controls | 4 months

SECONDARY OUTCOMES:
Booster effect on antibody titers against influenza 2009 H1N1 of 2010 Fluarix vaccination | February 2011

CONTACTS AND LOCATIONS:
Overall Officials: Vanda Friman, MD, Ph.D, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Transplant Institute, Sahlgrenska University Hospital, Gothenburg, Västra Götaland County, Sweden

REFERENCES:
- [Derived] Felldin M, Andersson B, Studahl M, Svennerholm B, Friman V. Antibody persistence 1 year after pandemic H1N1 2009 influenza vaccination and immunogenicity of subsequent seasonal influenza vaccine among adult organ transplant patients. Transpl Int. 2014 Feb;27(2):197-203. doi: 10.1111/tri.12237. Epub 2013 Dec 2. PMID 24289658